CLINICAL TRIAL: NCT04938765
Title: Randomized and Placebo Controlled Study to Evaluate the Effect of Magnesium Sulfate on Intraoperative Neuromonitoring.
Brief Title: Effect of Magnesium Sulfate Bolus on Intraoperative Neuromonitoring
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 5210244
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Intraoperative Neurophysiological Monitoring; Magnesium Sulfate
Keywords: multimodal analgesia
MeSH Terms: interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Intervention Model Description: Prospective double blind randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Study drug or the placebo will be administered after inducing general anesthesia hence patient will be masked. study drug or the placebo will be administered by the anesthesia team and this will not be disclosed to the neuro monitoring team who sits far away from the anesthesia workstation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Magnesium sulfate arm (Experimental): MgSo4 diluted to 20% will be administered at 40 mg/kg dosed to ideal body weight over 10min to the study arm followed by 10mg/kg/hr infusion.
  Interventions: Drug: Magnesium sulfate
- Normal Saline (Placebo Comparator): 20 ml of normal saline bolus will be administered to the control group over 10 mins.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Magnesium sulfate — Effect of 40mg/kg Magnesium sulfate bolus dosed to ideal body weight on intraoperative neuromonitoring
  Arms: Magnesium sulfate arm
Drug: Normal Saline — 20 ml of normal saline bolus will be administered to the control group over 10 mins.
  Arms: Normal Saline

SUMMARY:
Magnesium Sulfate(MgSo4) is increasingly being used as part of the multimodal pain regimen in the perioperative period. The intraoperative neurophysiological monitoring (IONM) is utilized in complex spine and cranial surgeries to assess the functional integrity of the neural pathways. The effect of Magnesium sulfate on IONM has not been studied.

This is a prospective, double blind, randomized placebo controlled trial to study the effect of Magnesium sulfate bolus on the amplitude and latency of somatosensory(SSEPs) and motor evoked potentials(MEPs) in patients undergoing surgery requiring IONM.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the effect of magnesium sulfate on the amplitude of the SSEP with tibial nerve stimulation. Secondary objectives are to study the effect of magnesium sulfate on the latency of SSEPs and the amplitude of MEPs in patients undergoing spine and/or cranial surgery requiring intraoperative neuromonitoring.

Background: Magnesium Sulfate is increasingly being used as part of the multimodal pain regimen in the perioperative period. The efficacy of intravenous (IV) magnesium sulfate in reducing the postoperative pain scores and/or postoperative opioid use has been established in several randomized controlled trials, systematic reviews, and meta-analyses. The multimodal intraoperative neurophysiological monitoring (IONM) is increasingly being utilized in complex spine surgeries to assess the functional integrity of the neural pathways. The goal of IONM is to avert permanent damage by proving real-time feedback from sensory tracts, motor tracts, and individual nerve roots thus alerting any impending injury which allows for modification of management in time.

Several factors like, hypoxia, hypercarbia, changes in blood pressure and temperature can affect the IONM in addition to direct surgical injury to neural structures. In addition, several drugs including anesthetic agents can have a significant effect on IONM. Hence anesthetic regimen is usually tailored to facilitate IONM during these surgeries. The infusion of propofol and remifentanil are commonly used for maintenance of anesthesia during these procedures. Opioid analgesics play a central role in the anesthetic cocktail as the pain associated with complex spinal surgery can be debilitating. However, opioids can also complicate the postoperative pain management by inducing opioid induced hyperalgesia and /or tolerance. The current trend is to implement a multimodal analgesic approach to achieve an additive or synergistic analgesic effect by targeting different receptors in the peripheral and central pain signaling pathways while minimizing opioid-related adverse effects. Magnesium sulfate has shown promising results when used as part of the multimodal pain management in previous studies in addition it can also has shown to attenuate the remifentanil-induced hyperalgesia which is commonly used as part of the anesthetic regimen. However, the effect of Magnesium Sulfate on intraoperative neuromonitoring is not been studied.

Methods Procedures involved (Research Interventions):

After obtaining the written informed consent and premedication, patients will be taken to the operating room. The standard ASA monitors will be applied. They will be monitored with electrocardiography, noninvasive and/or invasive blood pressure (BP), pulse oximetry, and temperature monitor along with brain function monitor to monitor the depth of anesthesia (Sedline monitor) during surgery.

After preoxygenation, the patient will be induced with general anesthesia using fentanyl 1-3 mg/kg or Remifentanil 1-3 mcg/kg, lidocaine 1-2 mg/kg, Propofol 1-3 mg/kg, and succinylcholine 1-2 mg/kg or Rocuronium 0.3-0.5 mg/kg. Inhalation anesthetic agents will not be used for induction or maintenance of anesthesia but may be used after the end of data collection for this study and/or during closing. Anesthetic infusion consisting of propofol 50-150 mg/kg, remifentanil 0.05-0.2 mg/kg will be started immediately after the induction for maintenance of general anesthesia and doses may be adjusted to higher amounts if needed. The BP will be maintained within 20% of patient's baseline using phenylephrine infusion or other appropriate vasoactive agents after the induction of anesthesia. End-tidal carbon dioxide will be maintained within normal limits. Patients will be actively warmed using a Bair Hugger™ or similar device(s) ("warmer(s)") to prevent any hypothermia.

In patients given rocuronium, neuromuscular blockage will be reversed before obtaining the baseline IONM recordings. The baseline set of SSEPs and MEPs will be recorded before the study drug administration and consisting of 2 to 4 measurements; T0 represents the average of these measurements. For study group, MgSo4 diluted to < 20% concentration in 20 ml normal saline will be administered as 40 mg/kg bolus dosed to ideal body weight over 10 min. For control group, 20 ml of normal saline bolus will be administered over 10 mins. Magnesium group will also be given continuous infusion of MgSO4 at 10mg/kg/hr. till the end of the surgery. Repeat SSEPs and MEPs will be recorded at the end of the bolus ("0" minutes) (T1) as well as 10 (T2) and 30 (T3) minutes following the completion of the bolus dose.

Patient's hemodynamic data also will be collected at baseline and every 5 mins up to 30 mins following the administration of the drug.

The T1,T2,T3 data will be compared with the To(baseline) data to evaluate the effect of MgSO4 on intraoperative neuromonitoring.

ELIGIBILITY:
Inclusion Criteria.

* Patients aged 18 to 80 years
* Belonging to American Society of Anesthesiologists physical status (ASA) I, II
* Undergoing elective spine or cranial surgery where intraoperative neuromonitoring including short latency somatosensory evoked potentials (SSEP or SEP) and transcranial electrical muscle motor evoked potentials recording from muscles (TceMEP or TcMEP or mMEP or MEP) is planned.

Exclusion Criteria:

* Magnesium use within the last 2 days, either intravenous or oral supplements.
* Patients with known electrolyte imbalances (Sodium <135 or >145 mmol/L OR Potassium < 3.5 or > 5.0 mmol/L, Magnesium >1.2 mmol/L.
* Severe cardiac or cardiac conduction disorders.
* Severe pulmonary disease.
* Patients with significant neuromuscular disorders or preexisting motor or sensory deficits other than focal upper limb neuropathy or focal cervical radiculopathy or mild cervical myelopathy.
* Severe Renal disease - serum creatinine of > 2 mg/dl.
* Pregnant or breastfeeding patients.
* Unable to obtain adequate baseline SSEPs and MEPs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in the amplitude of SSEPs. | Up to 30 minutes after the end of bolus dose of MgSO4 or Normal saline.
  Baseline SSEP recording is done before the administration of MgSo4 or placebo and will be compared with the SSEPs measured at 0,10 and 30 minutes following the end of the bolus dose of MgSO4 or normal saline. Any change in the amplitude will be analyzed. For SSEPs, 50% reduction in amplitude will be considered as significant change.

SECONDARY OUTCOMES:
Change in the latency of SSEP compared to baseline. | Up to 30 minutes after the end of bolus dose of MgSO4 or Normal saline.
  Baseline SSEP recording is done before the administration of MgSo4 or placebo and will be compared with the SSEPs measured at 0, 10 and 30 minutes following the end of the bolus dose of MgSO4 or normal saline.10% increase in latency will be considered as significant change.
Change in the amplitude of MEPs. | Up to 30 minutes after the end of bolus dose of MgSO4 or Normal saline.
  Baseline MEP recording is done before the administration of MgSo4 or placebo and will be compared with the MEPs measured at 0, 10 and 30 minutes following the end of the bolus dose of MgSO4 or normal saline. Any change in the amplitude of MEPs will be analyzed .For MEPs, 75% decrease in amplitude is considered as significant change

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Vandse, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albrecht E, Kirkham KR, Liu SS, Brull R. Peri-operative intravenous administration of magnesium sulphate and postoperative pain: a meta-analysis. Anaesthesia. 2013 Jan;68(1):79-90. doi: 10.1111/j.1365-2044.2012.07335.x. Epub 2012 Nov 1. PMID 23121612
- [Background] De Oliveira GS Jr, Castro-Alves LJ, Khan JH, McCarthy RJ. Perioperative systemic magnesium to minimize postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2013 Jul;119(1):178-90. doi: 10.1097/ALN.0b013e318297630d. PMID 23669270
- [Background] Guo BL, Lin Y, Hu W, Zhen CX, Bao-Cheng Z, Wu HH, Kaye AD, Duan JH, Qu Y. Effects of Systemic Magnesium on Post-operative Analgesia: Is the Current Evidence Strong Enough? Pain Physician. 2015 Sep-Oct;18(5):405-18. PMID 26431120
- [Background] Arumugam, S. , S. M. Lau, C. and Chamberlain, R. (2016) Perioperative Adjunct Magnesium Decreases Postoperative Opioid Requirements-A Meta-Analysis. International Journal of Clinical Medicine, 7, 297-308. doi: 10.4236/ijcm.2016.75032.
- [Background] Dehkordy ME, Tavanaei R, Younesi E, Khorasanizade S, Farsani HA, Oraee-Yazdani S. Effects of perioperative magnesium sulfate infusion on intraoperative blood loss and postoperative analgesia in patients undergoing posterior lumbar spinal fusion surgery: A randomized controlled trial. Clin Neurol Neurosurg. 2020 Sep;196:105983. doi: 10.1016/j.clineuro.2020.105983. Epub 2020 Jun 2. PMID 32521394
- [Background] Kizilcik N, Koner O. Magnesium Sulfate Reduced Opioid Consumption in Obese Patients Undergoing Sleeve Gastrectomy: a Prospective, Randomized Clinical Trial. Obes Surg. 2018 Sep;28(9):2783-2788. doi: 10.1007/s11695-018-3243-7. PMID 29754384
- [Background] Shin HJ, Kim EY, Na HS, Kim TK, Kim MH, Do SH. Magnesium sulphate attenuates acute postoperative pain and increased pain intensity after surgical injury in staged bilateral total knee arthroplasty: a randomized, double-blinded, placebo-controlled trial. Br J Anaesth. 2016 Oct;117(4):497-503. doi: 10.1093/bja/aew227. Epub 2016 Oct 17. PMID 28077538
- [Background] Ballesteros-Flores CG, Garrido-Aguirre E, Carrillo-Esper R, et al. Hypomagnesemia in the perioperative period. Current concepts. Rev Mex Anest. 2013;36(2):114-118.
- [Background] Whittaker JD, Downes F, Becker H, Garnham A, Wall M. Influence of Perioperative Serum Magnesium for Cardiac and Noncardiac Morbidity and Mortality Following Emergency Peripheral Vascular Surgery. J Cardiothorac Vasc Anesth. 2019 Feb;33(2):474-479. doi: 10.1053/j.jvca.2018.05.042. Epub 2018 May 28. PMID 30045811
- [Background] Herroeder S, Schonherr ME, De Hert SG, Hollmann MW. Magnesium--essentials for anesthesiologists. Anesthesiology. 2011 Apr;114(4):971-93. doi: 10.1097/ALN.0b013e318210483d. PMID 21364460
- [Background] Hicks MA, Tyagi A. Magnesium Sulfate. [Updated 2020 May 8]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2021 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK554553/
- [Background] Okusanya BO, Oladapo OT, Long Q, Lumbiganon P, Carroli G, Qureshi Z, Duley L, Souza JP, Gulmezoglu AM. Clinical pharmacokinetic properties of magnesium sulphate in women with pre-eclampsia and eclampsia. BJOG. 2016 Feb;123(3):356-66. doi: 10.1111/1471-0528.13753. Epub 2015 Nov 24. PMID 26599617
- [Background] Yanni DS, Ulkatan S, Deletis V, Barrenechea IJ, Sen C, Perin NI. Utility of neurophysiological monitoring using dorsal column mapping in intramedullary spinal cord surgery. J Neurosurg Spine. 2010 Jun;12(6):623-8. doi: 10.3171/2010.1.SPINE09112. PMID 20515347
- [Background] Huang ZF, Chen L, Yang JF, Deng YL, Sui WY, Yang JL. Multimodality Intraoperative Neuromonitoring in Severe Thoracic Deformity Posterior Vertebral Column Resection Correction. World Neurosurg. 2019 Jul;127:e416-e426. doi: 10.1016/j.wneu.2019.03.140. Epub 2019 Apr 11. PMID 30981802
- [Background] Minahan RE. Intraoperative neuromonitoring. Neurologist. 2002 Jul;8(4):209-26. doi: 10.1097/00127893-200207000-00001. PMID 12803681
- [Background] Cofano F, Zenga F, Mammi M, Altieri R, Marengo N, Ajello M, Pacca P, Melcarne A, Junemann C, Ducati A, Garbossa D. Intraoperative neurophysiological monitoring during spinal surgery: technical review in open and minimally invasive approaches. Neurosurg Rev. 2019 Jun;42(2):297-307. doi: 10.1007/s10143-017-0939-4. Epub 2018 Jan 8. PMID 29313181
- [Background] Sloan TB, Heyer EJ. Anesthesia for intraoperative neurophysiologic monitoring of the spinal cord. J Clin Neurophysiol. 2002 Oct;19(5):430-43. doi: 10.1097/00004691-200210000-00006. PMID 12477988
- [Background] Nunes RR, Bersot CDA, Garritano JG. Intraoperative neurophysiological monitoring in neuroanesthesia. Curr Opin Anaesthesiol. 2018 Oct;31(5):532-538. doi: 10.1097/ACO.0000000000000645. PMID 30020157
- [Background] Santonocito C, Noto A, Crimi C, Sanfilippo F. Remifentanil-induced postoperative hyperalgesia: current perspectives on mechanisms and therapeutic strategies. Local Reg Anesth. 2018 Apr 9;11:15-23. doi: 10.2147/LRA.S143618. eCollection 2018. PMID 29670398